CLINICAL TRIAL: NCT05701540
Title: A Multicenter, Double-blind, Randomized, Active-controlled Phase 4 Study to Evaluate the Efficacy and Safety of Tegoprazan in GERD Patients With Nighttime Heartburn
Brief Title: A Study to Evaluate the Efficacy and Safety of Tegoprazan in GERD Patients With Nighttime Heartburn
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IN_APA_403
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — tegoprazan; Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tegoprazan 50mg (Experimental): Tegoprazan 50mg, once daily, oral administration for two weeks
  Interventions: Drug: Tegoprazan
- Esomeprazole 40mg or 20mg (Active Comparator): 1. In case of ERD patients: Esomeprazole 40mg, qd, oral administration for two weeks
  2. In case of NERD patients: Esomeprazole 20mg, qd, oral administration for two weeks
  Interventions: Drug: Esomeprazole

INTERVENTIONS:
Drug: Tegoprazan — Tegoprazan 50mg tablet
  Arms: Tegoprazan 50mg
Drug: Esomeprazole — Esomeprazole 20mg tablet
  1. For patients with ERD: two Esomeprazole 20mg tablets
  2. For patients with NERD: one Esomeprazole 20mg tablet
  Arms: Esomeprazole 40mg or 20mg

SUMMARY:
This study aims to compare the nighttime heartburn improvement effect of Tegoprazan 50mg and Esomeprazole 40mg(or 20mg) in patients with GERD.

DETAILED DESCRIPTION:
This is a multi-center, double-blind, randomized, active-controlled phase 4 study. Subjects will be randomly assigned to one of the two treatment groups (tegoprazan 50mg, esomeprazole 40mg or 20mg).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged between 19 and 75 years
2. Subjects who have erosive reflux disease or non-erosive reflux disease

Exclusion Criteria:

1. Unable to undergo upper GI endoscopy
2. Symptoms of primary or secondary esophageal movement disorders
3. Subjects who have undergone or are scheduled to undergo surgery that can affect gastric acid secretion(e.g. upper gastrectomy, vagotomy, etc)

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Estimated)
Dates: Start 2023-03-24 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of days without nighttime heartburn during the 2-week dosing period | 2 weeks
  Percentage of days without nighttime heartburn = Number of days without nighttime heartburn symptoms during the dosing period / Number of days when nighttime heartburn was assessed x 100

SECONDARY OUTCOMES:
Time to first nighttime hearturn-free interval(days) | 2 weeks
  Number of days to reach the first day without symptoms of nighttime heartburn after the administration of investigational drug
Percentage of days without daytime heartburn during the 2-week dosing period | 2 weeks
  Percentage of days without daytime heartburn = Number of days without daytime heartburn symptoms during the dosing period / Number of days when daytime heartburn was assessed x 100

CONTACTS AND LOCATIONS:
Overall Officials: Sang Kil Lee, Ph.D, Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, South Korea